CLINICAL TRIAL: NCT06814353
Title: An International Multicenter Prospective Cohort Study Investigating the Intraoperatively Observed Site of Origin and Growth Pattern of the Molecular Groups of Medulloblastoma
Brief Title: Intraoperatively Observed Site of Origin and Growth Pattern of Medulloblastoma
Acronym: ISOP
Status: Enrolling by invitation | Type: Observational
Sponsor: Christian Dorfer (Other)
Collaborators: Medical University of Vienna (Other); University Hospital Tuebingen (Other); Utrecht University (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor-Investigator, Christian Dorfer, Assoc. Prof. Priv.-Doz. Dr. Christian Dorfer, MBA, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: ISOP (EK 1967/2023)
Record Dates: First submitted 2024-12-26; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Medulloblastoma
Keywords: Medulloblastoma
MeSH Terms: conditions — Medulloblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Tumor samples which are gained during surgery will be analyzed. Histopathologic and genetic classification data are obtained by immunohistochemistry for β-Catenin, Yap1, Gab1, p53 and complementary mutation analysis of the by DNA methylation profiling (Illumina, San Diego, California), which is the current gold standard for the allocation to the molecular group of medulloblastoma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- WNT-MB: Patients with a medulloblastoma of the subgroup MB, WNT(Wingless)-activated according to the WHO classification 2021.
  Interventions: Procedure: Intraoperative assessment of the site of origin and growth pattern
- SHH-MB: Patients with a medulloblastoma of the subgroup MB, SHH (Sonic Hedgehog)-activated according to the World Health Organization (WHO) classification 2021. This subgroup can be further differentiated into SHH-activated (SHH-MB) TP53-wildtype and MB, SHH-activated TP53-mutant.
  Interventions: Procedure: Intraoperative assessment of the site of origin and growth pattern
- Group 3 and Group 4: Patients with a medulloblastoma of the subgroup MB, non-WNT/non-SHH activated MB (Group 3 and 4) according to the WHO classification 2021.
  Interventions: Procedure: Intraoperative assessment of the site of origin and growth pattern

INTERVENTIONS:
Procedure: Intraoperative assessment of the site of origin and growth pattern — The assessment of the epicenter and extension and therefore the assumed origin of tumor growth is conducted by an experienced pediatric neurosurgeon blinded to group allocation based on the intraoperative impression. The anatomical features and site of origin are systematically documented on the surgical form in all cases of this study.
  Other Names: Assessment of the site and origin and growth pattern on preoperative MRI; Evaluation of anatomic features; Imaging feature extraction and characterization; Histopathological and molecular analysis

SUMMARY:
The goal of this observational study is to provide accurate and systematic data on the site of origin and growth pattern of medulloblastoma from a neurosurgical perspective. By integrating intraoperative, radiological and genetic classification data, this study will contribute to our current understanding of the development, site of origin and growth pattern of medulloblastoma and advance the predictive accuracy of radiogenomics models. Patients with histologically confirmed medulloblastoma who undergo surgical resection at a high-volume center with expertise in pediatric neurosurgery will be included.

The main questions it aims to answer are:

* Is there a significant difference between the intraoperatively observed site of origin and the preoperatively or postoperatively radiologically assessed site of origin of medulloblastoma?
* How does the intraoperatively observed site of origin align with the site of origin associated with the molecular group based on the developmental cell lineage concept of medulloblastoma?
* Does incorporating the intraoperatively observed site of origin as a feature improve the predictive accuracy of radiomic models for molecular group classification?

Participants will:

* Undergo intraoperative assessment of site of origin and growth pattern by an experienced pediatric neurosurgeon.
* Have their site of origin and growth pattern evaluated on pre- and postoperative magnetic resonance imaging by an neuroradiologist with expertise in pediatric brain tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are referred for surgical resection of a medulloblastoma at a hospital with expertise in pediatric neurooncology
* Both pediatric patients (aged < 18 years at the time of diagnosis) and adult patients (aged > 18 years at the time of diagnosis)

Exclusion Criteria:

* Patients who are preoperatively admitted with severe tumor hemorrhage accompanied by clinical deterioration are excluded because these patients frequently do not receive magnetic resonance imaging as would be necessary for the present study, and the intraoperative assessment of the STO is limited in accuracy due to decreased visibility caused by the intra- and extratumoral hemorrhage.
* If an intraoperative complication occurs (e.g. bleeding) which impairs visibility of the neuroanatomic structures and does not allow an accurate assessment of the STO, the patient is excluded.
* If the histopathological and molecular analysis does not confirm the diagnosis of a MB, the patient has to be excluded as well.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Both adult and pediatric patients who undergo surgical resection of a histologically confirmed medulloblastoma at a center with expertise in pediatric neurosurgery
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Rate of agreement between the intraoperatively observed site of origin and preoperatively radiologically assessed site of origin of medulloblastoma | From enrollment to the end of treatment at 6 weeks
  The intraoperatively observed site of origin is categorized into brainstem, cerebellar hemispheres and cerebellar vermis.The intraoperatively observed site of origin is assessed by an experienced pediatric neurosurgeon blinded to subgroup allocation and systemically documented in surgical forms.
  The location and site of origin is assessed by one expert neuroradiologist with expertise in pediatric brain tumor imaging who is blinded to the group allocation.
  Preoperative magnetic resonance imaging (MRI) includes at least T1-weighted, T2-weighted, fluid-attenuated inversion recovery (FLAIR) and contrast-enhanced, T1-weighted sequences. The presumed site of origin is analyzed following a simplification of the concept of Patay et al., 2015 with the following levels: posterior/posterolateral brainstem, midline vermis or cerebellar hemispheres based on the preoperative imaging aspect.
  The rate of agreement between both measures is reported.

SECONDARY OUTCOMES:
The rate of agreement between the intraoperatively observed site of origin and the site of origin presumably associated with a molecular group (standard of reference) based on the developmental cell lineage concept of medulloblastoma | From enrollment to the end of treatment at 6 weeks
  The intraoperatively observed site of origin is categorized into brainstem, cerebellar hemispheres and cerebellar vermis. The intraoperatively observed site of origin is assessed by an experienced pediatric neurosurgeon blinded to subgroup allocation and systemically documented in surgical forms.
  Histopathological and genetic data are used to identify the molecular subgroup of the MB.
  According to the current literature (Northcott et al., 2019), the site of origin presumably associated with the molecular group is categorized as brainstem for WNT-MB, the cerebellar hemisphere for SHH-MB and the cerebellar vermis for non-WNT/non-SHH-MB.
  The rate of agreement between the intraoperatively observed site of origin (brainstem, cerebellar hemisphere, cerebellar vermis) and the site of origin presumably associated with a molecular group (brainstem, cerebellar hemisphere, cerebellar vermis) is reported for each molecular group separately.
The neurological outcome measured as KPS scores stratified by the intraoperatively observed site of origin | From enrollment to the end of treatment at 6-weeks
  The intraoperatively observed site of origin is categorized into brainstem, cerebellar hemispheres and cerebellar vermis. The intraoperatively observed site of origin is assessed by an experienced pediatric neurosurgeon blinded to subgroup allocation and systemically documented in surgical forms.
  The neurological outcome at 6 weeks- follow-up is assessed using the Karnofsy Performance Scale.
  Patients are stratified by the intraoperatively observed site of origin into three groups (brainstem, cerebellar hemispheres, cerebellar vermis).
  The KPS scores are reported as boxplots with median and interquartile range for the three groups separately.
Predictive accuracy of radiogenomic models | From enrollment to the end of treatment at 6 weeks
  For construction of nomograms, the entire study sample will be split into a training cohort (TC) and a validation cohort (VC) in the ratio 7:3. Independent binary nomograms will be developed for each of the 4 subgroups. Receiver operating characteristics (ROC) curves will be generated following application of individual subgroup-specific nomograms to assign scores for patients in the TC. The methodology will be repeated in the VC. Optimal cutoff of total scores for individual subgroup-specific nomograms will be generated from the ROC curves from the TC for acceptable range of specificity and sensitivity, and their applicability was subsequently tested in the VC. Area under the curve (AUC) with 95% CI will be used for interpretation and reporting. MRI-based nomograms will be constructed two times, with the intraopely observed site of origin being the only additional feature. AUCs with 95% CI will be compared among the nomograms.

CONTACTS AND LOCATIONS:
Locations (4):
- Department of Neurosurgery, Medical University of Vienna, Vienna, Vienna, Austria
- Germany (2):
  - Department of Neurosurgery, Charité Berlin, Berlin
  - Section of Pediatric Neurosurgery, University Hospital of Tuebingen, Tübingen
- Department of Neurosurgery, Princess Maxima Centre for Pediatric Oncology, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided